CLINICAL TRIAL: NCT06934941
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of NM-101
Brief Title: Phase 1 Single Ascending Dose Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neuramedy Co. Ltd. (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: NM-101-01; NM-101 (Other: Neuramedy)
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects
Keywords: Single Ascending Dose study

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NM-101 (Experimental): NM-101 iv
  Interventions: Drug: NM-101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NM-101 — NM-101 IV versus placebo
  Other Names: Placebo
  Arms: NM-101
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Phase 1, double-blind, placebo-controlled, single-centre, single ascending dose escalation study to assess safety and tolerability of a monoclonal antibody, NM-101 in healthy volunteer subject and multiple system atrophy (MSA) patients.

DETAILED DESCRIPTION:
Phase 1, double-blind, placebo-controlled, single-centre, single ascending dose escalation study to assess safety and tolerability of a monoclonal antibody, NM-101 in healthy volunteer subject and multiple system atrophy (MSA) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male Healthy subjects, 18 to 60 years of age and in good health with no clinically significant abnormality identified on the medical history, physical examination or laboratory evaluation at screening
2. Body weight≥ 45kg and body mass index between 18 - 30 kg/m2
3. Normal blood pressure (systolic >90 and <140 mmHg, diastolic >40 and <90mmHg) and pulse rate 40-100bpm at screening visit. Blood pressure and pulse are measured after 3 minutes in supine position
4. Baseline QTc must be <450msec for men and <470msec for women
5. Normal 12-lead electrocardiogram at screening
6. No clinically significant abnormal laboratory test values at screening
7. No clinically significant findings on the clinical neurological and ophthalmic examinations at screening and at baseline
8. Good venous access in both arms
9. Willing to consent to participate in study prior to study specific screening procedures with the understanding that the subject has the right to withdraw from the study at any time without prejudice
10. Female subject who is surgically sterile, is postmenopausal, or agrees to use a highly effective method of birth control (2 methods strongly recommended) during the study and for 6 months after the dosing of NM-101.

Exclusion Criteria:

1. History of serious adverse reaction or hypersensitivity to biological agents including immunoglobulins
2. Presence or history of any allergy requiring acute or chronic treatment; seasonal allergic rhinitis can be permitted unless the subject is taking systemic medication (nasal spray or local treatments permitted). Subjects having clinically significant drug or food allergies are also excluded.
3. History of autoimmune or inflammatory disease
4. Clinically significant (i.e., active) cardiovascular disease (e.g., hypertension, arrhythmia, myocardial infarction, heart failure, long QT syndrome or other conditions causing prolongation of the QT/QT interval corrected with Fridericia's formula [QTcF]) prior to screening.
5. History of cerebral vascular accident or stroke. Subjects having high risk of developing a stroke are also excluded.
6. History or positive test results at screening for human immunodeficiency virus (HIV), hepatitis B, hepatitis C
7. Positive in tuberculosis screening test (Quantiferon test)
8. Active infection within 4 weeks from screening and body temperature >38℃
9. Active immunization within 3 months prior to dosing of NM-101
10. History or clinically significant evidence of cardiovascular, endocrine (e.g. diabetes mellitus), respiratory, renal, hepatic, gastrointestinal, haematological neurologic, psychiatric or other disease
11. Chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary track
12. History or presence of malignancy including solid tumors and hematologic malignancies except for basal cell and squamous cell carcinoma of the skin that had been completely excised and were considered cured with no evidence of disease ≥ 3 years
13. Participation in a clinical study during the previous 24 weeks i.e. from completion of the previous study to the planned first administration of the current study
14. Loss of >500mL blood including blood donation within 12 weeks prior to screening visit
15. Intake more than 24 units of alcohol per week (1 unit=250mL of beer, 100mL of wine or 35mL of spirits)
16. Smokers >5 cigarettes or the equivalent in tobacco daily. Must have been willing to abstain from using tobacco and tobacco-containing products for 72 hours prior to the dosing of NM-101 and during the inpatient monitoring period.
17. Treatment with any prescription medication and/or over-the-counter products (excluding acetaminophen, hormone replacement therapy (HRT) and birth control) within 30 days prior to dosing of NM-101. Routine vitamin therapy is allowed.
18. History of drug or alcohol abuse within the past 5 years, a positive urine drug test and/or a positive alcohol urine test at Screening visit
19. Surgery other than minor cosmetic surgery and minor dental surgery within 3 months from the screening visit
20. History of lumbar surgery for any reasons (e.g., herniated disc) or other contraindications to having al lumbar puncture (LP)
21. Vigorous physical exercise 48 hours prior to screening
22. Women with a positive pregnancy test at screening
23. Women who are breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
To determine the pharmacokinetic profile of NM-101 after a single iv infusion | Pre-dose, 0, 0.5, 1, 2, 4, 6, 8, 12hour post-dose at Day 1 and Day 2, 3, 4, 8, 15, 22, 29 and week 6, 8, 12
  Peak plasma drug concentration (Cmax)
To determine the pharmacokinetic profile of NM-101 after a single iv infusion | Pre-dose, 0, 0.5, 1, 2, 4, 6, 8, 12hour post-dose at Day 1 and Day 2, 3, 4, 8, 15, 22, 29 and week 6, 8, 12
  Area under the plasma concentration versus time curve (AUC) at steady-state and until last observation
To determine the pharmacokinetic profile of NM-101 after a single iv infusion | Pre-dose, 0, 0.5, 1, 2, 4, 6, 8, 12hour post-dose at Day 1 and Day 2, 3, 4, 8, 15, 22, 29 and week 6, 8, 12
  Concentration at trough
To determine the pharmacokinetic profile of NM-101 after a single iv infusion | Pre-dose, 0, 0.5, 1, 2, 4, 6, 8, 12hour post-dose at Day 1 and Day 2, 3, 4, 8, 15, 22, 29 and week 6, 8, 12
  Time to maximum drug concentration
To determine the pharmacokinetic profile of NM-101 after a single iv infusion | Pre-dose, 0, 0.5, 1, 2, 4, 6, 8, 12hour post-dose at Day 1 and Day 2, 3, 4, 8, 15, 22, 29 and week 6, 8, 12
  half-life of drug
To determine the pharmacokinetic profile of NM-101 after a single iv infusion | Pre-dose, 0, 0.5, 1, 2, 4, 6, 8, 12hour post-dose at Day 1 and Day 2, 3, 4, 8, 15, 22, 29 and week 6, 8, 12
  Volume distribution of drug
To determine the pharmacokinetic profile of NM-101 after a single iv infusion | Pre-dose, 0, 0.5, 1, 2, 4, 6, 8, 12hour post-dose at Day 1 and Day 2, 3, 4, 8, 15, 22, 29 and week 6, 8, 12
  Clearance rate of drug

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided